CLINICAL TRIAL: NCT07221565
Title: ImmuneNet: Quantum-Synaptic Immunotherapy Mapping
Brief Title: Quantum-Synaptic Immunotherapy Mapping Using Low-Frequency Electromagnetic Resonance and Machine Learning-Based Cytokine Forecasting
Acronym: QSIT
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Truway Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TWH-QSIT-IMMUNENET-2025-01
Record Dates: First submitted 2025-10-23; First posted 2025-10-28 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Systemic Lupus Erythematosus; Rheumatoid Arthritis; Multiple Sclerosis; Autoimmune Diseases; Chronic Inflammatory Syndromes; Immune Dysregulation
Keywords: Quantum Immunotherapy; Electromagnetic Resonance Therapy; Low-Frequency Electromagnetic Fields; Immune Cell Synchronization; Cytokine Forecasting; AI-Driven Immunomodulation; Truway Health ClinicalChain; Non-pharmacologic Immune Regulation; Autoimmune Flare Reduction; Machine Learning in Immunology
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid; Multiple Sclerosis; Autoimmune Diseases | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to receive either active low-frequency electromagnetic resonance therapy or sham stimulation. Each arm follows the same 12-week schedule. Outcomes are compared across parallel groups to evaluate immune-regulation effects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind trial. Devices are pre-coded by an independent technician so that neither participants nor investigators can distinguish active from sham units. Outcomes assessors remain blinded until database lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active Low-Frequency Electromagnetic Resonance (LF-EMR) (Experimental): Participants in the experimental arm will receive non-invasive low-frequency electromagnetic resonance (LF-EMR) therapy three times per week for twelve weeks. Each session uses a calibrated emitter producing resonant fields between 7-40 Hz at amplitudes below 2 microtesla. The treatment is designed to promote synchronized signaling among immune effector cells and reduce autoimmune flare frequency.
  Interventions: Device: Low-Frequency Electromagnetic Resonance Therapy (LF-EMR); Device: Sham Resonance Device (Inactive Control); Drug: Low-Dose Naltrexone (LDN)
- Sham Electromagnetic Stimulation (Placebo Control) (Sham Comparator): Participants in the control arm will undergo identical procedures with a deactivated (sham) LF-EMR device that emits no measurable electromagnetic field. This arm controls for placebo and procedural effects. Neither participants nor investigators will know which device is active or inactive.
  Interventions: Device: Low-Frequency Electromagnetic Resonance Therapy (LF-EMR); Device: Sham Resonance Device (Inactive Control); Drug: Low-Dose Naltrexone (LDN)

INTERVENTIONS:
Device: Low-Frequency Electromagnetic Resonance Therapy (LF-EMR) — A non-invasive medical device that generates low-frequency electromagnetic fields (7-40 Hz < 2 μT) targeted at harmonizing immune-cell electromagnetic communication. Participants receive 20-minute sessions three times weekly for twelve weeks. The device is cleared for investigational use under Truway Health protocol TWH-QSIT-IMMUNENET-2025-01.
  Other Names: Quantum-Synaptic Resonance Device (QSR-01)
Device: Sham Resonance Device (Inactive Control) — A visually identical device programmed to remain inactive and emit no electromagnetic field. Used to maintain blinding and assess placebo response. Participants follow the same treatment schedule as the active group.
  Other Names: Placebo LF-EMR Unit
Drug: Low-Dose Naltrexone (LDN) — Participants assigned to this adjunct pharmacologic arm will receive low-dose naltrexone (4.5 mg oral capsule once daily at bedtime) for twelve weeks.
  Low-dose naltrexone is hypothesized to reduce pro-inflammatory cytokine activity and enhance endogenous endorphin-mediated immune regulation. The dose is well below the standard 50 mg level used for addiction therapy and has been studied for autoimmune and inflammatory disorders.
  This arm will allow assessment of potential synergy between electromagnetic-resonance signaling and pharmacologic immune modulation.
  Manufacturer / Source:
  Compounded formulation supplied by Truway Health Clinical Pharmacy, New York, NY (cGMP-certified).
  Route of Administration:
  Oral (capsule)
  Dosage Form:
  Capsule, 4.5 mg
  Frequency / Duration:
  Once daily for 12 weeks
  Intended Use:
  Investigational immune-modulating therapy to complement non-pharmacologic intervention.
  Other Names: Naltrexone Hydrochloride, 4.5 mg oral capsule

SUMMARY:
The ImmuneNet study is a Phase I/II clinical trial sponsored by Truway Health, Inc. It will test whether gentle, low-frequency electromagnetic resonance (LF-EMR) can influence how immune cells communicate and synchronize with each other. The goal is to see if this "quantum-synaptic" signaling effect can help stabilize immune activity and reduce the number of autoimmune flare-ups in people living with conditions such as lupus, rheumatoid arthritis, or multiple sclerosis.

Participants will receive either an active or a sham (placebo) LF-EMR session three times per week for twelve weeks. Each session is completely non-invasive. Blood samples will be collected to study cytokines (immune-system messenger molecules), gene-expression patterns, and electrical field coherence among immune cells.

A machine-learning system will analyze these data to predict inflammation patterns and guide individualized treatment settings. All participant data will be securely recorded and time-stamped to ensure transparency and privacy.

The expected outcome of the study is a measurable reduction in autoimmune flare frequency and symptom severity, along with improved understanding of how electromagnetic signaling might safely regulate immune function.

DETAILED DESCRIPTION:
This exploratory, randomized, double-blind, parallel-assignment Phase I/II trial is designed to evaluate the safety, tolerability, and biological activity of low-frequency electromagnetic resonance (LF-EMR) for immune modulation.

Rationale and Objectives Autoimmune diseases involve abnormal immune signaling that leads to chronic inflammation. Emerging biophysical evidence suggests that immune cells generate and respond to ultra-low-frequency electromagnetic fields that may coordinate cytokine release and cell communication. The ImmuneNet protocol seeks to harness this phenomenon through controlled, resonant electromagnetic exposure to promote immune homeostasis.

Methods Approximately 120 adults aged 18-70 with stable autoimmune disease will be enrolled at Truway Health Research Centers in New York, NY and Austin, TX. Participants will be randomly assigned in a 1:1 ratio to active or sham LF-EMR stimulation. Active participants will receive 7-40 Hz resonant fields (< 2 microtesla) for 20 minutes per session, three times weekly for twelve weeks. Sham participants will undergo identical procedures with the device inactive.

Blood samples collected at baseline, week 6, week 12, and six-month follow-up will undergo multiplex cytokine analysis, RNA sequencing, and electrophysiologic coherence mapping. Machine-learning models will be trained to forecast cytokine cascades and flare probability.

Outcome Measures The primary endpoint is reduction in documented autoimmune flare frequency over six months. Secondary endpoints include changes in serum cytokine synchronization index, transcriptomic shift magnitude, patient-reported global health scores, and adverse-event incidence.

Ethics and Oversight The study will follow Good Clinical Practice (GCP) guidelines and be reviewed by an independent institutional review board. Participation is voluntary, and informed consent will be obtained from all subjects.

Expected Impact If successful, the trial will demonstrate a safe, non-pharmacologic approach to immune regulation and establish a data framework for future AI-guided quantum-resonant therapies. The knowledge gained could lead to new treatment options for autoimmune and chronic inflammatory diseases while reducing reliance on long-term immunosuppressive drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18-70 years.
2. Clinical diagnosis of a systemic autoimmune disorder (e.g., systemic lupus erythematosus, rheumatoid arthritis, or multiple sclerosis) confirmed for at least 12 months.
3. Stable disease-modifying therapy or corticosteroid regimen for at least 8 weeks prior to enrollment.
4. Willingness to maintain current medication schedule for the duration of the study.
5. Ability to provide written informed consent and comply with study procedures.
6. Access to stable internet or smartphone connection for digital consent verification and symptom tracking.

Exclusion Criteria:

1. Presence of an implanted medical or electronic device (e.g., pacemaker, defibrillator, deep brain stimulator).
2. Pregnancy or lactation.
3. Active infection, malignancy, or significant hepatic, renal, or cardiovascular disease.
4. Known photosensitivity, seizure disorder, or history of uncontrolled epilepsy.
5. Prior participation in any electromagnetic or quantum resonance study within the past 6 months.
6. Use of biologic or investigational therapy initiated within the previous 3 months.
7. Inability to attend at least 80% of treatment sessions or follow-up visits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2034-10-23 (Estimated); Study Completion 2034-10-23 (Estimated)

PRIMARY OUTCOMES:
Change in Autoimmune Flare Frequency | Baseline to Month 6
  Number of clinically confirmed autoimmune flare events during the 6-month observation period compared to baseline, using validated disease-specific scoring systems (e.g., SLEDAI for lupus, DAS-28 for rheumatoid arthritis, or EDSS for multiple sclerosis).

SECONDARY OUTCOMES:
Cytokine Synchronization Index (CSI) | Baseline, Week 12, and Month 6
  Change in cytokine synchronization index (CSI) calculated from multiplex cytokine panels (IL-6, TNF-α, IFN-γ, IL-10) using Fourier-transformed oscillatory coherence values between cytokine pairs.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Solomon, President & CEO, Principal Investigator — Truway Health, Inc.
Locations (1):
- Truway Health, Inc. www.truwayhealth.com (401 E 34th Street, S11P, New York, NY 10016), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available for secondary research analyses following publication of primary results. Shared data will include participant-level demographics, clinical outcomes, cytokine panels, and RNA sequencing results.
  Data will be accessible via the Truway Health ClinicalChain Data Repository, a blockchain-secured storage and access system ensuring traceable data integrity and compliance with HIPAA and GDPR standards.
  Access requests may be submitted to Truway Health, Inc. (help@truwayhealth.com) and will be reviewed by the sponsor's Data Access Committee. Researchers must provide a data use proposal and agree to a data-sharing agreement.
  IPD will become available approximately 12 months after study completion and remain available for a minimum of 5 years following initial publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months post-study completion
Access Criteria: Proposal review by Truway Health Data Access Committee; data-sharing agreement required
URL: https://www.truwayhealth.com

REFERENCES:
- See also: Truway Health Official Website — https://www.truwayhealth.com
- Available data/document: Study Protocol: IPD — https://www.truwayhealth.com — The Truway Health ClinicalChain repository will host de-identified datasets, full study protocol, and statistical analysis plan following publication. Access will be provided through blockchain-verified credentials to ensure compliance and auditability.